CLINICAL TRIAL: NCT00875290
Title: Gerber Pump Trial: Effectiveness of Continuous Subcutaneous Insulin Infusion (CSII) and Real-Time Sensor Augmentation (RTSA) in 0-3 Years Old Diabetes Patients; A One Year Randomized Controlled Clinical Trial.
Brief Title: The Effectiveness of Continuous Glucose Monitoring in Diabetes Treatment for Infants and Young Children
Acronym: Gerber RTSA
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seattle Children's Hospital (Other)
Collaborators: The Gerber Foundation (Other); Medtronic (Industry)
Responsible Party: Patricia Fechner, M.D., Seattle Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GerberPumpStudy
Record Dates: First submitted 2009-04-02; First posted 2009-04-03 (Estimated); Last update posted 2011-08-05 (Estimated); Status verified 2011-08

CONDITIONS: Diabetes Mellitus, Type I
Keywords: Diabetes Mellitus, Type I; Children; Insulin pump therapy; Continuous glucose monitor
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): Observational arm
- Real-time glucose sensor (Experimental): Subjects wear real-time glucose sensor
  Interventions: Device: Real-time glucose sensor

INTERVENTIONS:
Device: Real-time glucose sensor — Children assigned to this intervention will use a real-time sensor continuously
  Other Names: Minimed Paradigm Real-time sensor
  Arms: Real-time glucose sensor

SUMMARY:
The purpose of this study is to see if the use of a real-time glucose sensor improves diabetes control in young children (less than 4 years old) with Type I diabetes when they are initiated on insulin pump therapy.

DETAILED DESCRIPTION:
A randomized controlled clinical trial involving patients 0-3 yrs old with type 1 diabetes. After successful screening the subjects will be randomized into one of two groups: a CSII group alone and a CSII group + Real Time Sensor Augmentation group (RTSA) group. The CSII group will serve as the control for the CSII+RTSA group. The trial will last for one year.

ELIGIBILITY:
Inclusion Criteria:

* Children less than 4 years of age with Type I diabetes for at least 3 months

Exclusion Criteria:

* Children greater than 4 years of age
* Monogenic diabetes

Ages: 3 Months to 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2008-11; Primary Completion 2014-11 (Estimated); Study Completion 2014-11 (Estimated)

PRIMARY OUTCOMES:
Reduce blood glucose variability among 0-3 year old children with type I diabetes. | 1 year

SECONDARY OUTCOMES:
Number of adverse events | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Fechner, MD, Principal Investigator — Seattle Children's Hospital
Locations (1):
- Seattle Children's Hospital, Seattle, Washington, United States